CLINICAL TRIAL: NCT02459938
Title: A Randomized Open-label Crossover Study to Compare the Safety and Efficacy of ZP-Glucagon to Injectable Glucagon in the Treatment of Insulin-induced Hypoglycemia in Subjects With Type-1 Diabetes
Brief Title: Safety and Efficacy of ZP-Glucagon to Injectable Glucagon for Hypoglycemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zosano Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CP-2014-004
Record Dates: First submitted 2015-05-21; First posted 2015-06-02 (Estimated); Last update posted 2016-08-16 (Estimated); Status verified 2016-08

CONDITIONS: Hypoglycemia
MeSH Terms: conditions — Hypoglycemia | interventions — Glucagon; Glucagon-Like Peptide 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- ZP-Glucagon 0.5 mg (Experimental): glucagon applied to the ZP transdermal microneedle patch system at a dose of 0.5 mg applied by means of a purpose built reusable applicator and worn for 30 minutes
  Interventions: Drug: Glucagon (ZP-Glucagon)
- ZP-Glucagon 1.0 mg (Experimental): glucagon applied to the ZP transdermal microneedle patch system at a dose of 1.0 mg applied by means of a purpose built reusable applicator and worn for 30 minutes
  Interventions: Drug: Glucagon (ZP-Glucagon)
- Glucagon by injection, 0.5 mg (Active Comparator): glucagon applied as GlucaGen (NovoNordisk) injector system at a dose of 0.5 mg
  Interventions: Drug: Glucagon (GlucaGen)
- Glucagon by injection, 1.0 mg (Active Comparator): glucagon applied as GlucaGen (NovoNordisk) injector system at a dose of 0.5 mg
  Interventions: Drug: Glucagon (GlucaGen)

INTERVENTIONS:
Drug: Glucagon (ZP-Glucagon) — chemically synthesized glucagon as delivered via transdermal microneedle patch system for 30 minutes
  Other Names: glucagon
  Arms: ZP-Glucagon 0.5 mg; ZP-Glucagon 1.0 mg
Drug: Glucagon (GlucaGen) — recombinant glucagon administered via subcutaneous injection
  Other Names: glucagon
  Arms: Glucagon by injection, 0.5 mg; Glucagon by injection, 1.0 mg

SUMMARY:
The purpose of this study is to determine whether glucagon administered by microneedle patch is comparable to glucagon administered by injection pen in the treatment of insulin-induced hypoglycemia.

DETAILED DESCRIPTION:
The purpose of this study is to compare ZP-Glucagon transdermal patch system at doses of 0.5 mg and 1 mg to glucagon by injection at doses of 0.5 mg and 1 mg by means of a 4 way crossover open label design. Eligible subjects giving informed consent will be randomised to a treatment sequence of each of the four treatments in one week intervals. At each treatment visit, subjects will undergo an insulin induction procedure designed to safely induce hypoglycemia, and then have a treatment applied, either by injection or by patch, and then monitored for return to normoglycemia.

ELIGIBILITY:
Inclusion Criteria:

* Women or men 18 to 60 years with type-1 diabetes on daily insulin treatment (basal-bolus injection regimen or insulin pump) for at least two years, on a total daily dose that has been stable for the last 3 months preceding enrollment (no more than 20% variation), and with a current level of glycated hemoglobin between 6.5% and 10%

Exclusion Criteria:

* Any history of hypoglycemic coma or hypoglycemic seizures.
* Any episode of severe hypoglycemia (requiring treatment) within one month prior to study start.
* Any history of pheochromocytoma or insulinoma

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2015-01; Primary Completion 2015-08 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects achieving normoglycemia | 30 minutes

SECONDARY OUTCOMES:
Time at which normoglycemia is first reached | 3 hours
Time at which maximal glucose levels are reached | 3 hours
Increases in blood glucose by 15 minute intervals | 3 hours
Peak Plasma Concentration (Cmax) | 3 hours
Area under the plasma concentration versus time curve (AUC) | 3 hours

CONTACTS AND LOCATIONS:
Overall Officials: Neale Cohen, MD, Principal Investigator — Baker ID Heart and Diabetes Institute
Locations (1):
- Nucleus Network, Melbourne, Victoria, Australia